CLINICAL TRIAL: NCT00177918
Title: Prospective Evaluations of Infectious Complications in Lung Transplant Recipients
Brief Title: Prospective Evaluations of Infectious Complication in Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, EJ Kwak, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY20040282
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Disorder Related to Lung Transplantation; Bronchiolitis Obliterans
Keywords: Lung Transplant
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers will be removed and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. All samples that are provided to outside facilities will be sent with a code number. Samples may be sent to other investigators not associated with this study to perform diagnostic testing (e.g., viral, fungal, bacterial and immunological). All samples will be provided to investigators not associated with the study without any identifiers and only contain a code number. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung transplant patients

SUMMARY:
The primary aim of this study is to determine prospectively the viral and C. pneumoniae infection prevalence and outcomes of infections in lung transplant recipients. The study will also determine the correlation of C. pneumoniae infection with the development of obliterans in lung transplant recipients.

DETAILED DESCRIPTION:
This is a prospective cohort study of lung transplant recipients and those who will undergo lung transplantation. Patients will be identified by the pulmonologist performing the bronchoscopy. The patient's sera (obtained from a one time blood draw of 10 milliliters - two tablespoons) and cell pellet of BAL will be frozen at -70º C. Once the active or non- OB status is determined by the pathologist, stored BAL fluid (cell pellet) will be analyzed. C.pneumoniae serum titers will also be measured and compared with stored pre-transplant sera. Left over cell pellet of the BAL fluid will be used to measure the presence of C. pneumoniae by PCR method. Additionally PCR will be performed for other viruses (CMV, EBV, HHV6 & 7, human metapneumo virus and human rhino virus). In addition, during the bronchoscopy procedure as part of the patient's standard of care, a biopsy is obtained. This is done during the bronchoscopy procedure. The tissue is then sent to the pathology lab. We will collect residual (excess) tissue samples to perform research related testing. This testing will determine if we can predict other types of infections and early onset of rejection. These determinations will assist clinicians in administering appropriate dosage levels of antibiotics required to prevent or treat infections and help stop the rejection process. The subject will be asked a few questions about pulmonary symptoms that will not take more than five minutes by one of the investigators or study coordinator. The subject's medical record will be reviewed for demographic information (age, sex, and race), lab results (standard to post transplant care), medication information, as well as any testing/procedures during the transplant follow-up period. This information and results of the tests/procedures will become part of the research record.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone lung transplantation or will undergo a lung transplant at the University of Pittsburgh Medical Center and are alive following transplant period will be eligible for the study.

Exclusion Criteria:

* Subjects not willing to participate in the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all lung transplant patients transplanted at UPMC
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2006-08 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
long term outcome after lung transplantation | five year follow up
  looking at death rate five years post lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: EJ Kwak, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States